CLINICAL TRIAL: NCT03505710
Title: A Phase 2, Multicenter, Open-Label, 2-Cohort Study of Trastuzumab Deruxtecan (DS-8201a), an Anti-HER2 Antibody Drug Conjugate (ADC), for HER2-Over-Expressing or -Mutated, Unresectable and/or Metastatic Non Small Cell Lung Cancer (NSCLC) (DESTINY-Lung01)
Brief Title: DS-8201a in Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing or -Mutated Non-Small Cell Lung Cancer
Acronym: DESTINY-Lung01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Last participant transitioned to alternative study.
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U204; 2017-004781-94 (EudraCT Number); JapicCTI-183916 (Registry Identifier: JAPIC)
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: HER2 over-expression; HER2 mutation; Unresectable or metastatic; Non-squamous; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: HER2 Overexpressing (Experimental): Participants with HER2-overexpressing(immunohistochemistry [IHC] 3+ or IHC 2+), unresectable and/or metastatic NSCLC adenocarcinoma who received 6.4 mg/kg trastuzumab deruxtecan (DS-8201a).
  Interventions: Drug: Trastuzumab deruxtecan
- Cohort 1a: HER2 Overexpressing (Experimental): Participants with HER2-overexpressing (immunohistochemistry [IHC] 3+ or IHC 2+), unresectable and/or metastatic NSCLC adenocarcinoma who received 5.4 mg/kg trastuzumab deruxtecan (DS-8201a).
  Interventions: Drug: Trastuzumab deruxtecan
- Cohort 2: HER2 Mutated (Experimental): Participants with HER2-mutated, unresectable and/or metastatic NSCLC who received 6.4 mg/kg trastuzumab deruxtecan (DS-8201a).
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Antibody component covalently conjugated to a drug component, prepared by dilution based on body weight for intravenous (IV) infusion.
  Other Names: DS-8201a; Experimental product

SUMMARY:
The primary objective of this trial is to evaluate the efficacy of trastuzumab deruxtecan in HER2-overexpressing and/or HER2-mutated advanced NSCLC participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old in Japan, ≥18 years old in other countries
* Pathologically documented unresectable and/or metastatic non-squamous NSCLC
* Has relapsed from or is refractory to standard treatment or for which no standard treatment is available
* For Cohort 1 and Cohort 1a: HER2-overexpression (IHC 2+ or 3+) status must be assessed and confirmed by Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory or equivalent, from an archival tumor tissue sample
* For Cohort 2 only: Participant has any known documented activating HER2 mutation from an archival tumor tissue sample analyzed by CLIA laboratory or equivalent. Note: HER2 mutation documented only from a liquid biopsy sample cannot be used for enrollment.
* Presence of at least 1 measurable lesion assessed by the investigator and based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Is willing and able to provide an adequate archival tumor tissue sample
* Is willing to undergo a tissue biopsy, after the completion of the most recent treatment regimen
* Has Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1

Exclusion Criteria:

* Had been previously treated with HER2-targeted therapies, except for pan-HER class tyrosine kinase inhibitors
* For Cohort 1 and Cohort 1a: Has known HER2 mutation
* Has a medical history of myocardial infarction, symptomatic congestive heart failure (CHF) (NYHA classes II-IV), unstable angina or serious cardiac arrhythmia
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out due to imaging at screening
* Has a QT interval corrected by Fridericia's formula (QTcF) prolongation to > 450 millisecond (ms) in males and > 470 ms in females
* Has a medical history of clinically significant lung disease
* Is suspected to have certain other protocol-defined diseases based on imaging at screening period
* Has history of any disease, metastatic condition, drug/medication use or other condition that might, per protocol or in the opinion of the investigator, compromise:

  1. safety or well-being of the participant or offspring
  2. safety of study staff
  3. analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (21):
- United States (9):
  - University of California San Diego (UCSD), La Jolla, California
  - University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine at St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Washington, Seattle, Washington
- France (5):
  - Centre Leon Berard, Lyon, Rhne
  - Hôpital Nord - CHU Marseille, Marseille
  - CHU Larrey, Toulouse
  - Hôpital Larrey, CHU-Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Shizuoka Cancer Center, Nakatogari, Sunto-gun
  - National Cancer Center Hospital, Chuo Ku, Tokyo
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Smit EF. Trastuzumab deruxtecan in HER2-mutant non-small-cell lung cancer: a plain language summary of the DESTINY-Lung01 study. Future Oncol. 2024;20(27):1961-1971. doi: 10.1080/14796694.2024.2355724. Epub 2024 Jul 16. PMID 39012221
- [Derived] Smit EF, Felip E, Uprety D, Nagasaka M, Nakagawa K, Paz-Ares Rodriguez L, Pacheco JM, Li BT, Planchard D, Baik C, Goto Y, Murakami H, Saltos A, Pereira K, Taguchi A, Cheng Y, Yan Q, Feng W, Tsuchihashi Z, Janne PA. Trastuzumab deruxtecan in patients with metastatic non-small-cell lung cancer (DESTINY-Lung01): primary results of the HER2-overexpressing cohorts from a single-arm, phase 2 trial. Lancet Oncol. 2024 Apr;25(4):439-454. doi: 10.1016/S1470-2045(24)00064-0. PMID 38547891
- [Derived] Li BT, Smit EF, Goto Y, Nakagawa K, Udagawa H, Mazieres J, Nagasaka M, Bazhenova L, Saltos AN, Felip E, Pacheco JM, Perol M, Paz-Ares L, Saxena K, Shiga R, Cheng Y, Acharyya S, Vitazka P, Shahidi J, Planchard D, Janne PA; DESTINY-Lung01 Trial Investigators. Trastuzumab Deruxtecan in HER2-Mutant Non-Small-Cell Lung Cancer. N Engl J Med. 2022 Jan 20;386(3):241-251. doi: 10.1056/NEJMoa2112431. Epub 2021 Sep 18. PMID 34534430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 181 participants were enrolled and treated at clinic centers in Japan, United States, France, Netherlands, and Spain.
Pre-assignment Details: Duration of follow-up (months) was defined as ((last visit date - enrollment date + 1)/365.25) × 12. Last visit date was the date of last clinical visit for ongoing participants, date of death for participants who died, or the last known contact date in survival follow-up for other participants who discontinued study drug.
Groups:
- Cohort 2: HER2 Mutated: Participants with HER2-mutated, unresectable and/or metastatic NSCLC to who received 6.4 mg/kg trastuzumab deruxtecan (DS-8201a).
  Trastuzumab deruxtecan: Antibody component covalently conjugated to a drug component, prepared by dilution based on body weight for intravenous (IV) infusion.
Period: Overall Study
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Started | 49 | 41 | 91
Completed (Study was Completed as last participant transitioned to alternative study) | 0 | 0 | 0
Not Completed | 49 | 41 | 91
Not completed — Progressive Disease | 24 | 17 | 43
Not completed — Clinical Progression | 6 | 8 | 3
Not completed — Adverse Event | 12 | 6 | 28
Not completed — Withdrawal by Subject | 1 | 3 | 7
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Death | 4 | 5 | 6
Not completed — Other Reasons | 1 | 1 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated | Total
Number analyzed (Participants) | 49 | 41 | 91 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 55 | 109
  >=65 years | 22 | 14 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (9.58) | 60.3 (10.22) | 60.3 (11.94) | 60.8 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 60 | 98
  Male | 30 | 22 | 31 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 13 | 4 | 31 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 1 | 7
  White | 31 | 31 | 40 | 102
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 19 | 23
Region of Enrollment [Number; unit: participants]
  Netherlands | 10 | 8 | 13 | 31
  United States | 19 | 13 | 35 | 67
  Japan | 12 | 3 | 23 | 38
  France | 0 | 3 | 15 | 18
  Spain | 8 | 14 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Independent Central Review Following Treatment With DS8201a in Participants With HER2-Over-Expressing or -Mutated Non-Small-Cell Lung Cancer (NSCLC)
Description: The Objective Response Rate (ORR) was the defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by independent central review (ICR) committee based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on ICR is reported.
Time Frame: From screening, up to 36 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 03 December 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Number analyzed (Participants) | 49 | 41 | 91
Percentage of Participants | 26.5 [15.0 to 41.1] | 34.1 [16.1 to 45.5] | 54.9 [44.2 to 65.4]

2. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Investigator Assessment Following Treatment With DS8201a in Participants With HER2-Over-Expressing or -Mutated Non-Small-Cell Lung Cancer (NSCLC)
Description: The Objective Response Rate (ORR) was defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigator assessment based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on investigator assessment is reported.
Time Frame: From screening, up to 36 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 03 May 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Number analyzed (Participants) | 49 | 41 | 91
Percentage of Participants | 28.6 [16.6 to 43.3] | 31.7 [18.1 to 48.1] | 61.5 [50.8 to 71.6]

3. Secondary Outcome: Duration of Response (DoR) Following Treatment With DS8201a in Participants With HER2-Over-Expressing or -Mutated Non-Small-Cell Lung Cancer (NSCLC)
Description: Duration of Response (DoR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR in participants with confirmed CR/PR based on independent central review and investigator assessment is reported.
Time Frame: From screening to documented tumor progression or death from any cause, up to 36 months (data cut-off)
Population: Duration of Response (DoR) was assessed in the Full Analysis Set of participants with confirmed CR/PR at data cut-off date of 03 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Number analyzed (Participants) | 13 | 12 | 50
months
  Independent Central Review | 5.8 [4.3 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 4.7 [4.0 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 9.3 [5.7 to 14.7]
  Investigator Assessment: number analyzed (Participants) | 11 | 3 | 30
  Investigator Assessment | 5.8 [4.7 to 11.3] | 7.0 [4.2 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 11.7 [7.2 to 16.9]

4. Secondary Outcome: Progression-Free Survival (PFS) Following Treatment With DS8201a in Participants With HER2-Over-Expressing or -Mutated Non-Small-Cell Lung Cancer (NSCLC)
Description: Progression-free survival (PFS) was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. PFS based on independent central review and investigator assessment is reported.
Time Frame: From date of enrollment to first objective radiographic tumor progression or death from any cause,, up to 36 months (data cut-off)
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 03 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Number analyzed (Participants) | 49 | 41 | 91
months
  Independent Central Review | 5.7 [2.8 to 7.2] | 6.7 [4.5 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 8.2 [6.0 to 11.9]
  Investigator Assessment | 5.7 [3.8 to 7.2] | 7.2 [4.1 to 8.4] | 9.3 [7.1 to 14.0]

5. Secondary Outcome: Overall Survival (OS) Following Treatment With DS8201a in Participants With HER2-Over-Expressing or -Mutated Non-Small-Cell Lung Cancer (NSCLC)
Description: Overall survival (OS) was defined as the time from the date of first dose of study drug to the date of death due to any cause.
Time Frame: From date of enrollment to death from any cause, up to 36 months (data cut-off)
Population: Overall survival (OS) was assessed in the Full Analysis Set at data cut-off date of 03 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Number analyzed (Participants) | 49 | 41 | 91
months | 12.4 [7.8 to 17.2] | NA [6.7 to NA] — Median OS and upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 17.8 [13.8 to 22.1]

6. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR) Following Treatment With DS8201a in Participants With HER2-Over-Expressing or -Mutated Non-Small-Cell Lung Cancer (NSCLC)
Description: Disease Control Rate (DCR) was defined as the percentage of participants who achieved a best overall response of CR, PR, or stable disease (SD) during study treatment. Confirmation of CR/PR was required. DCR based on independent central review and investigator assessment is reported.
Time Frame: From first dose, up to 36 months (data cut-off)
Population: Disease control rate was assessed in the Full Analysis Set at data cut-off date of 03 May 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
Number analyzed (Participants) | 49 | 41 | 91
Percentage of Participants
  Independent Central Review | 68.9 [53.4 to 81.8] | 77.5 [61.6 to 89.2] | 93.0 [85.4 to 97.4]
  Investigator Assessment | 75.5 [61.1 to 86.7] | 78.0 [62.4 to 89.4] | 94.5 [87.6 to 98.2]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 47 days after last dose of the study drug, up 36 months.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug.
Arm/Group | Cohort 1: HER2 Overexpressing | Cohort 1a: HER2 Overexpressing | Cohort 2: HER2 Mutated
All-Cause Mortality (participants affected / at risk) | 42/49 | 32/41 | 72/91
Serious Adverse Events (participants affected / at risk) | 28/49 | 18/41 | 40/91
Other Adverse Events (participants affected / at risk) | 46/49 | 41/41 | 91/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HER2 Overexpressing (N=49) | Cohort 1a: HER2 Overexpressing (N=41) | Cohort 2: HER2 Mutated (N=91)
Disease Progression (General disorders) | 6 | 4 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 7
Pneumonia (Infections and infestations) | 4 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3
Seizure (Nervous system disorders) | 1 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Central Nervous System Necrosis (Nervous system disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Covid-19 Pneumonia (Infections and infestations) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Duodenal Stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1
Oesophageal Infection (Infections and infestations) | 1 | 0 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 | 0 | 1
Partial Seizures (Nervous system disorders) | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Radiation Necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 1
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Troponin I Increased (Investigations) | 0 | 0 | 1
Troponin Increased (Investigations) | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Disease Complication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: HER2 Overexpressing (N=49) | Cohort 1a: HER2 Overexpressing (N=41) | Cohort 2: HER2 Mutated (N=91)
Nausea (Gastrointestinal disorders) | 28 | 30 | 69
Diarrhoea (Gastrointestinal disorders) | 13 | 14 | 39
Vomiting (Gastrointestinal disorders) | 14 | 13 | 42
Constipation (Gastrointestinal disorders) | 15 | 10 | 36
Abdominal Pain (Gastrointestinal disorders) | 2 | 5 | 8
Stomatitis (Gastrointestinal disorders) | 6 | 3 | 6
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 8
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0 | 5
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 7
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 5
Neutrophil Count Decreased (Investigations) | 11 | 2 | 28
White Blood Cell Count Decreased (Investigations) | 6 | 2 | 18
Lymphocyte Count Decreased (Investigations) | 6 | 2 | 13
Weight Decreased (Investigations) | 12 | 8 | 22
Alanine Aminotransferase Increased (Investigations) | 5 | 4 | 14
Aspartate Aminotransferase Increased (Investigations) | 6 | 4 | 17
Platelet Count Decreased (Investigations) | 8 | 3 | 12
Blood Creatinine Increased (Investigations) | 5 | 3 | 5
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 1 | 6
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 7
Fatigue (Gastrointestinal disorders) | 16 | 20 | 30
Asthenia (General disorders) | 6 | 7 | 16
Malaise (General disorders) | 9 | 3 | 13
Pyrexia (General disorders) | 1 | 3 | 16
Oedema Peripheral (General disorders) | 2 | 5 | 14
Non-Cardiac Chest Pain (General disorders) | 3 | 5 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 22 | 19 | 32
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 4 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 18
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 5 | 42
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 6
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Anaemia (Blood and lymphatic system disorders) | 15 | 13 | 33
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 8
Dizziness (Nervous system disorders) | 10 | 3 | 8
Headache (Nervous system disorders) | 4 | 5 | 16
Dysgeusia (Nervous system disorders) | 4 | 3 | 13
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 7
Muscluar Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Pneumonia (Infections and infestations) | 5 | 2 | 18
Urinary Tract Infection (Infections and infestations) | 3 | 2 | 9
Insomnia (Psychiatric disorders) | 2 | 0 | 12
Anxiety (Psychiatric disorders) | 1 | 3 | 8
Depression (Psychiatric disorders) | 0 | 0 | 5
Dry Eye (Eye disorders) | 0 | 3 | 8
Hypertension (Vascular disorders) | 0 | 0 | 7
Hypotension (Vascular disorders) | 4 | 0 | 7
Weight Increased (Investigations) | 0 | 3 | 4
Fatigue (General disorders) | 16 | 21 | 30
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03505710/Prot_SAP_000.pdf